CLINICAL TRIAL: NCT01449747
Title: Mechanism of Reduced Response to DPP-4 Inhibitor in Patients With Type 2 Diabetes Mellitus
Brief Title: Pharmacokinetics Study of Dipeptidyl Peptidase 4 Inhibitor to Control Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ji Hyun Kim, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCENDO-01
Record Dates: First submitted 2011-09-29; First posted 2011-10-10 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Dipeptidyl peptidase IV inhibitors; Glucagon-like peptide 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Active Comparator): sitagliptin hypo-response patients
  Interventions: Drug: Sitagliptin
- control group (Sham Comparator): sitagliptin response patients
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin (100mg, per oral) once a day.
  Other Names: Januvia

SUMMARY:
The purpose of this study is to confirm the mechanism of reduced response to DPP-4 inhibitor in some patients with type 2 diabetes and evaluate appropriate patients to treat with DPP-4 inhibitor

DETAILED DESCRIPTION:
Sitagliptin, a DPP-4 inhibitor was used as an incretin enhancer in clinical practice first. In clinical trials, sitagliptin showed effective control of blood glucose level in type 2 diabetes and 100 mg once daily with metformin was similar to sulfonylurea (glipizide) with metformin in lowering HbA1c. Mostly in practice, stable blood glucose levels were maintained after change of sulfonylurea to sitagliptin in type 2 diabetes treatment. However, in some cases, there were abrupt severe hyperglycemia and uncontrolled blood glucose level after drug change to sitagliptin.

Several mechanism could be considered for reduced response to DPP-4 inhibitor in some type 2 diabetes patients. Firstly, significantly reduced secretion of glucagon-like peptide 1 (GLP-1) more than expected in diabetes or functional defect of GLP-1 activity could be the mechanism of loss of GLP-1 effect irrespective of DPP-4. Secondly, mutation or functional defect of DPP-4 enzyme could not be inhibited by DPP-4 inhibitor. Thirdly, GLP-1 receptor mutation or other defect in β-cell responsiveness to GLP-1 leads to reduction of response to DPP-4 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with less than 15 yrs of disease duration
* BMI between 22-27 kg/m2
* HbA1c ≤ 9% at recruitment

  1. Study group

After change sulfonylurea to sitagliptin in case of metformin and sulfonylurea therapy

1. Increase of fasting blood glucose over 20 mg/dL or postprandial glucose over 30 mg/dL within several days or
2. Increase of HbA1c over 1% within 2-3 months without abrupt increase of blood glucose levels within several days

   * Sulfonylurea dose : less than glimepiride 4mg or gliclazide 120mg or glibenclamide 10mg
   * Metformin dose : 500~2000mg
3. Reduced response to sitagliptin should be made a decision by investigators after understanding the condition of patients surely.

2. Control group

* Age, sex, BMI matched patients with same condition of study patients
* After change sulfonylurea to sitagliptin in case of metformin plus sulfonylurea therapy, no change of blood glucose levels like above or stable HbA1c change within 1% within 2-3 months

Exclusion Criteria:

* Other causes of increase of blood glucose levels except drug change
* Patients with history of insulin treatment
* Patients taking thiazolidinediones, alpha-glucosidase inhibitors, GLP-1 analogue or DPP-4 inhibitors
* Patients with renal, hepatic dysfunction
* Patients with diabetic complications such as coronary heart disease, cerebrovascular disease, proliferative diabetic retinopathy or diabetic gastroparesis
* Patients taking medications affecting glucose level

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hyun Kim, Dr, Principal Investigator — The Catholic University of Korea
Locations (2):
- South Korea (2):
  - The Catholic University of Korea; St.Paul's Hospital, Seoul
  - The Catholic University of Korea; Seoul St. Mary's Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-responder: Sitagliptin non-response patients
- Responder: Sitagliptin response patients
Period: Overall Study
Arm/Group | Non-responder | Responder
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-responder | Responder | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (5.7) | 57.4 (7.0) | 58.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 9 | 18
Duration of diabetes mellitus [Mean (Standard Deviation); unit: years] | 7.2 (5.5) | 5.2 (2.7) | 6.2 (4.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (1.7) | 24.4 (3.8) | 24.8 (2.9)
HbA1c [Mean (Standard Deviation); unit: %] | 7.7 (0.6) | 6.6 (0.7) | 7.2 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Active Glucagon-like Peptide 1 (GLP-1) Before and After Sitagliptin Treatment
Description: Plasma concentrations of active GLP-1 were measured at 0, 15, 30, 45, 60, 90, 120 and 180 min during the meal tolerance test (MTT). Second measurement of active GLP-1 were measured with MTT after taking sitagliptin 100 mg 1 hour before the test.
Time Frame: 0, 15, 30, 45, 60, 90, 120, 180 min pre and post-dose
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 12 | 12
pmol/L
  baseline 0 min | 7.0 (6.6) | 6.1 (1.9)
  baseline 15 min | 10.6 (8.0) | 14.1 (24.4)
  baseline 30 min | 15.7 (10.3) | 14.3 (20.2)
  baseline 45 min | 14.7 (8.2) | 9.3 (4.3)
  baseline 60 min | 13.7 (6.8) | 8.4 (2.7)
  baseline 90 min | 10.6 (5.4) | 7.6 (2.1)
  baseline 120 min | 11.3 (6.8) | 7.4 (2.1)
  baseline 180 min | 12.6 (8.7) | 7.1 (2.5)
  post-dose 0 min | 13.6 (9.4) | 10.5 (4.5)
  post-dose 15 min | 24.0 (16.0) | 26.0 (39.9)
  post-dose 30 min | 28.4 (11.0) | 34.3 (53.1)
  post-dose 45 min | 22.4 (11.3) | 27.1 (37.6)
  post-dose 60 min | 21.7 (11.3) | 22.8 (27.1)
  post-dose 90 min | 19.3 (10.8) | 16.5 (7.6)
  post-dose 120 min | 22.0 (10.8) | 16.4 (6.5)
  post-dose 180 min | 20.5 (8.3) | 13.5 (7.0)

2. Secondary Outcome: Differences of DPP-4 Activity After Sitagliptin Treatment Between Responder and Non-responder Groups
Description: The DPP-4 activity was measured at baseline and 0, 15, 30, 45 and 60 min during the meal tolerance test. Second measurement of DPP-4 activity was measured with MTT after taking sitagliptin 100 mg 1 hour before the test. Plasma DPP-4 activity during meal tolerance test is expressed as percentage activity relative to baseline. DPP-4 activity % was calculated using the following formula : (DPP-4 activity at time t / Baseline DPP-4 activity) × 100.
Time Frame: 0, 15, 30, 45, 60 min post-dose
Measure: Mean (Standard Deviation); unit: percentage of DPP4 activity
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 12 | 12
percentage of DPP4 activity
  baseline | 100 (0) | 100 (0)
  Sitagliptin 0 min | 67.2 (13.2) | 40.5 (9.9)
  Sitagliptin 15 min | 67.3 (18.6) | 39.2 (11.2)
  Sitagliptin 30 min | 67.7 (13.1) | 38.7 (9.2)
  Sitagliptin 45 min | 59.6 (18.7) | 33.5 (8.4)
  Sitagliptin 60 min | 58.5 (12.5) | 44.3 (7.7)

3. Primary Outcome: Plasma Concentration of Total GLP-1 Before and After Sitagliptin Treatment
Description: Plasma concentrations of total GLP-1 were measured at 0, 15, 30, 45, 60, 90, 120 and 180 min during the meal tolerance test. Second measurement of total GLP-1 were measured with MTT after taking sitagliptin 100 mg 1 hour before the test.
Time Frame: 0, 15, 30, 45, 60, 90, 120, 180 min pre and post-dose
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 12 | 12
pmol/L
  baseline 0 min | 25.6 (26.9) | 15.6 (16.2)
  baseline 15 min | 30.5 (26.1) | 20.4 (19.7)
  baseline 30 min | 36.2 (26.8) | 22.4 (17.0)
  baseline 45 min | 30.9 (18.9) | 25.5 (21.0)
  baseline 60 min | 31.8 (20.9) | 21.7 (19.9)
  baseline 90 min | 31.8 (24.3) | 19.2 (17.1)
  baseline 120 min | 31.3 (22.2) | 19.9 (18.0)
  baseline 180 min | 34.5 (28.3) | 19.3 (17.5)
  post-dose 0 min | 23.0 (27.8) | 16.4 (17.6)
  post-dose 15 min | 28.4 (27.9) | 20.6 (20.7)
  post-dose 30 min | 26.3 (19.4) | 20.6 (18.1)
  post-dose 45 min | 29.2 (27.2) | 18.9 (18.3)
  post-dose 60 min | 26.5 (29.1) | 18.6 (19.2)
  post-dose 90 min | 26.2 (30.1) | 18.1 (17.0)
  post-dose 120 min | 26.7 (30.5) | 18.7 (16.1)
  post-dose 180 min | 26.0 (25.8) | 18.2 (18.2)

4. Primary Outcome: Plasma Concentration of Total Glucose-dependent Insulinotropic Polypeptide (GIP) Before and After Sitagliptin Treatment
Description: Plasma concentrations of total GIP were measured at 0, 15, 30, 45, 60, 90, 120 and 180 min during the meal tolerance test. Second measurement of total GIP were measured with MTT after taking sitagliptin 100 mg 1 hour before the test.
Time Frame: 0, 15, 30, 45, 60, 90, 120, 180 min pre and post-dose
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 12 | 12
pmol/L
  baseline 0 min | 13.8 (4.5) | 12.3 (6.9)
  baseline 15 min | 42.3 (30.7) | 40.3 (28.1)
  baseline 30 min | 109.6 (49.9) | 60.2 (39.8)
  baseline 45 min | 109.6 (43.5) | 54.1 (37.9)
  baseline 60 min | 83.0 (22.6) | 52.0 (37.7)
  baseline 90 min | 66.3 (22.6) | 44.7 (25.5)
  baseline 120 min | 61.7 (27.9) | 39.0 (23.9)
  baseline 180 min | 39.9 (17.9) | 30.0 (18.2)
  post-dose 0 min | 10.5 (4.0) | 10.3 (5.3)
  post-dose 15 min | 34.2 (14.0) | 26.3 (15.6)
  post-dose 30 min | 90.8 (34.7) | 33.1 (23.5)
  post-dose 45 min | 77.6 (37.8) | 38.5 (23.5)
  post-dose 60 min | 61.5 (26.1) | 37.7 (25.4)
  post-dose 90 min | 44.2 (15.7) | 38.2 (41.6)
  post-dose 120 min | 43.8 (15.3) | 35.0 (39.0)
  post-dose 180 min | 32.8 (9.2) | 24.7 (25.6)

5. Primary Outcome: Change in AUC of Active GLP-1, Total GLP-1 and Total GIP Between Before and After Sitagliptin Treatment
Description: Plasma concentrations of active GLP-1, total GLP-1 and total GIP were measured at 0, 15, 30, 45, 60, 90, 120 and 180 min during the meal tolerance test. Second measurements were measured with MTT after taking sitagliptin 100 mg 1 hour before the test. Comparisons were made using Area under the curve (AUC) values and incremental area under the curve (ΔAUC) of active GLP-1, total GLP-1 and total GIP before and after the addition of sitagliptin.
Time Frame: 0, 15, 30, 45, 60, 90, 120, 180 min pre and post-dose
Measure: Mean (Standard Deviation); unit: pmol*min/L
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 12 | 12
pmol*min/L
  baseline AUC active GLP-1 | 2181.7 (1099.6) | 1578.2 (807.5)
  baseline AUC total GLP-1 | 5766.5 (4229.7) | 3680.2 (3209.3)
  baseline AUC total GIP | 10216.7 (4226.1) | 7575.6 (4608.3)
  post-dose AUC active GLP-1 | 3898.5 (1547.5) | 3535.1 (2769.1)
  post-dose AUC total GLP-1 | 4794.5 (4949.8) | 3373.6 (3169.8)
  post-dose AUC total GIP | 8784.6 (2449.2) | 5929.4 (4711.2)
  ΔAUC active GLP-1 | 1716.8 (1350.7) | 1956.8 (2910.7)
  ΔAUC total GLP-1 | -972.0 (1030.4) | -306.7 (883.6)
  ΔAUC total GIP | -1432.1 (2738.0) | -1646.2 (1817.7)

ADVERSE EVENTS:
Arm/Group | Non-responder | Responder
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No